CLINICAL TRIAL: NCT02218463
Title: Treatment of Prepubertal Labial Adhesions: A Prospective Comparison of Topical Emollient Versus Topical Estrogen.
Brief Title: Treatment of Prepubertal Labial Adhesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Missouri, Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMH14010039
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Prepubertal Labial Adhesions
Keywords: Vulvar disease, adhesions, topical therapy; Labial adhesions prepubertal girls; Labial agglutination; Labial fusion
MeSH Terms: conditions — Vulvar Diseases; Tissue Adhesions | interventions — Estradiol; cetyl alcohol, propylene glycol, sodium lauryl sulfate non-lipid cleansing lotion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cetaphil (Active Comparator): Apply a pea-sized amount to the labial adhesion with lateral traction twice daily
  Interventions: Drug: Cetaphil
- Estradiol Cream 0.01% (Active Comparator): Apply a pea-sized amount to the labial adhesion with lateral traction twice daily
  Interventions: Drug: Estradiol cream 0.01%

INTERVENTIONS:
Drug: Estradiol cream 0.01% — Apply a pea-sized amount to the labial adhesion with lateral traction twice daily
  Other Names: Estrace Vaginal
  Arms: Estradiol Cream 0.01%
Drug: Cetaphil — Apply a pea-sized amount to the labial adhesion with lateral traction twice daily
  Arms: Cetaphil

SUMMARY:
First-line treatment for labial adhesions in prepubertal girls has been topical estrogen. This study aims to evaluate an alternative and less costly option of treatment with potentially less side effects.

Primary Hypothesis:

There will be a difference in complete resolution of labial adhesions with topical estrogen with lateral traction as compared to an emollient with lateral traction.

DETAILED DESCRIPTION:
The etiology of labial adhesions is unclear but appears to be related to hypoestrogenism in combination with vulvar irritation. For many years, first-line treatment for labial adhesions in prepubertal girls has been topical estrogen. With the use of topical estrogen, 50% of labial adhesions resolve in 2 to 3 weeks and most labial adhesions resolve with 6 weeks of treatment. However, because topical estrogen is systemically absorbed, its use is associated with side effects such as breast budding, vulvar hyperpigmentation, vaginal bleeding. There is a high risk of recurrence of labial adhesions of up to 35% after treatment with topical estrogen. In addition, topical estrogen is costly. Therefore, there continues to be controversy over the optimal treatment of labial adhesions in prepubertal girls.

Generally, for medical treatment of labial adhesions, topical estrogen is applied to the adhesion whist applying gentle lateral traction to promote separation of the labia. It is, therefore, plausible that the lateral traction applied to the adhesion site is what ultimately results in the separation of the labial fusion, while the use of estrogen improves healing after mechanical separation.

This is a single site, prospective, randomized, double-blinded study evaluating the comparative effectiveness of topical estrogen with lateral traction versus topical emollient with lateral traction for the treatment of labial adhesions in prepubertal girls.

ELIGIBILITY:
Inclusion Criteria:

* Prepubertal girls ages 3 months to 12 years with labial adhesions

Exclusion Criteria:

* Presence of underlying dermatologic conditions such as lichen sclerosis, severe atopic dermatitis, psoriasis or vitiligo
* Presence of systemic conditions that can have vulvar manifestations such as Crohn's disease and Behçet disease
* Presence of disorders requiring immunosuppressant treatment
* Previous surgical separation of labial adhesions

Ages: 3 Months to 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tazim Dowlut-McElroy, MD, Principal Investigator — University of Missouri, Kansas City; Julie L Strickland, MD, MPH, Study Director — University of Missouri-Kansas City; Children's Mercy Hospital
Locations (1):
- Children's Mercy Hospitals & Clinics, Kansas City, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cetaphil | Estradiol Cream 0.01%
Started | 21 | 22
Completed | 18 | 19
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetaphil | Estradiol Cream 0.01% | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Full Range); unit: months] | 33 [5 to 84] | 26 [4 to 108] | 29 [4 to 108]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 22 | 43
% introital closure [Number; unit: participants]
  25% | 1 | 0 | 1
  50% | 5 | 4 | 9
  75% | 4 | 7 | 11
  100% | 11 | 11 | 22
Thickness of labial adhesion [Count of Participants; unit: Participants]
  Thin | 5 | 4 | 9
  Intermediate | 14 | 17 | 31
  Thick | 2 | 1 | 3
Urinary tract infection [Count of Participants; unit: Participants]
  Present | 0 | 2 | 2
  Absent | 21 | 20 | 41
Vulvovaginitis [Count of Participants; unit: Participants]
  Present | 0 | 0 | 0
  Absent | 21 | 22 | 43
Pain with activity [Count of Participants; unit: Participants]
  Present | 1 | 1 | 2
  Absent | 20 | 21 | 41
Postvoid dribbling [Count of Participants; unit: Participants]
  Present | 1 | 0 | 1
  Absent | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Complete Resolution of Labial Adhesion.
Description: The first assessment will be 3 weeks after initiation of treatment. The final assessment will be 6 weeks after initiation of treatment.
Time Frame: 3 weeks and 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cetaphil | Estradiol Cream 0.01%
Number analyzed (Participants) | 21 | 22
Participants | 21 | 22
Statistical Analysis 1: Comparison: Cetaphil vs Estradiol Cream 0.01%; Assessment of complete resolution between the 2 study arms; Test type: Superiority; p = 0.206, Fisher Exact

2. Secondary Outcome: Composite Severity Scale of Labial Adhesion Over Time
Description: Response to treatment of labial adhesion is dependent not only upon the size of the adhesion but also the thickness. A more accurate measurement of response to treatment would, therefore, incorporate both measurements. For this study, the percentage of closure of the introitus at presentation was assigned an ordinal value as follows: 1=25%, 2=50%, 3=75%, and 4=100%. The degree of thickness of the labial adhesion was also measured in a similar fashion: 1=thin, 2=intermediate and 3= thick. Those that were resolved received a rating of 0 on both scales. A composite severity scale was created by multiplying the value assigned to the percentage of introital closure by that assigned to the thickness of the adhesion for each of the 3 study visits. The composite severity scale ranged from 0 to 12. This allowed a comparison of treatment effect between each group over time wherein a lower composite severity score corresponded to a less severe labial adhesion.
Time Frame: 3 weeks and 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cetaphil | Estradiol Cream 0.01%
Number analyzed (Participants) | 21 | 22
units on a scale
  Baseline | 6.3 (3.1) | 6.2 (2.0)
  3 weeks | 2.3 (2.4) | 1.5 (1.7)
  6 weeks | 1.9 (2.1) | 1.6 (1.9)
Statistical Analysis 1: Comparison: Cetaphil vs Estradiol Cream 0.01%; Time Effect; Test type: Superiority; p = 0.0001, ANOVA
Statistical Analysis 2: Comparison: Cetaphil vs Estradiol Cream 0.01%; Treatment Effect; Test type: Superiority; p = 0.370, ANOVA
Statistical Analysis 3: Comparison: Cetaphil vs Estradiol Cream 0.01%; Treatment by time interaction; Test type: Superiority; p = 0.425, ANOVA

ADVERSE EVENTS:
Arm/Group | Cetaphil | Estradiol Cream 0.01%
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 1/21 | 1/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetaphil (N=21) | Estradiol Cream 0.01% (N=22)
Vulvar irritation (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No